CLINICAL TRIAL: NCT06844552
Title: Low Frequency High Intensity- Pulsed Magnetic Fields (LF-HI-PEMF) in Pain and Inlfammation
Brief Title: Diamagnetic Therapy in Pain and Inflammation
Acronym: DiaPI
Status: Recruiting | Type: Observational
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Luca Gallelli, Clinical Professor, University of Catanzaro
Other Study IDs: PEMFs
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Pain; Inflammation
MeSH Terms: conditions — Pain; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Treated: Low Frequency High Intensity- Pulsed Magnetic Fields - LF-HI-PEMF
- Treated + topical treatment: Low Frequency High Intensity- Pulsed Magnetic Fields - LF-HI-PEMF plus topical treatment + topical treatment
- topical treatment: topical treatment

SUMMARY:
This is a prospective longitudinal single-center clinical study on pain patients treated with Low Frequency High Intensity- Pulsed Magnetic Fields (LF-HI-PEMF; diamagnetic therapy) . Patients were enrolled at baseline (T0) and then were monitored at 30 days (T1), 60 days (T2), 90 days (T3). and 360 days (T4). The first efficacy end-point was the statistically significant difference (P<0.05) in VAS scale between T2-T4 and T0.

DETAILED DESCRIPTION:
This is a prospective longitudinal single-center clinical study on pain patients treated with Low Frequency High Intensity- Pulsed Magnetic Fields (LF-HI-PEMF; diamagnetic therapy) at the Pain Medicine Room of the Clinical Pharmacology and Pharmacovigilance Operative Unit of the "Renato Dulbecco" University Hospital of Catanzaro. Patients were enrolled at baseline (T0) and then were monitored during the follow-up (T1; 1 months; T2; 2 months; T3; 3 months; T4: 1 year). At the beginning of the study, all enrolled patients signed the informed consent before admission to the study. After the enrollment (T0) and during the follow ups (T1-T4), clinical and laboratory data were collected directly by the medical staff involved in the study and Zung SAS, Zung SDS and SF-36 questionnaires were administered. The dedicated database evaluated and recorded any systemic or local side effects. The Low Frequency High Intensity- Pulsed Magnetic Fields - LF-HI-PEMF was locally used. In patients that experienced low efficacy, a topical treatment was added. A group of patients that refused PEMFs or without indication for PEMFs, a topical treatment was used. Before the admission to this study, all the enrolled patients received systemic treatments without clinical benefit. The first efficacy end-point was the statistically significant difference (P<0.05) in VAS scale between T1 and T0, T2 and T1 and between T3 and T2-T0 and and T4 vs T3,T2,T1,T0

* the statistically significant difference (P<0.05) in functional mobility and walking ability (six minutes walking test) between T2 and T0 and between T3 and T2
* the statistically significant difference (P<0.05) in mood disorders (Zung SAS and Zung SDS) between T2 and T0 and between T3 and T2

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes between 18 and 75 years old
2. Patients with pain and or inflammation (e.g. osteoarthritis, trauma, prostatitis)
3. Patients with VAS (Visual Analogue Scale) intensities higher than 5/10 who did not respond to systemic medication therapy.
4. Patients who can comprehend the study's objectives and adhere to the clinical instructions, return for follow-up, and complete the evaluation questionnaires.
5. Patients able to provide their written informed consent to participate to the study and to use their data anonymously for scientific purposes

Exclusion Criteria:

1. presence of active malignancy of any type or history of malignancy
2. Local or systemic infection.
3. Uncooperative patient or suffering from neurological disorders, therefore unable to follow the clinical instructions or unable to provide informed consent for participation in the study or who have not provided written consent.
4. Any case not described in the inclusion criteria. Patients with contraindication to magnetic resonance imaging

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After the enrollment (T0) and during the follow ups (T1-T3), clinical and laboratory data were collected directly by the medical staff involved in the study and Zung SAS, Zung SDS questionnaires were administered. The dedicated database evaluated and recorded any systemic or local side effects. At the beginning of the study (T0) low Frequency High Intensity- Pulsed Magnetic Fields - LF-HI-PEMF was topically used in agreement with leaflet of the instrument with or without topical treatment. A group of patients received a treatment with topical compounds in agreement with the leaflet. Before the admission to this study, all the enrolled patients received systemic treatments without clinical benefit
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-07-19 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
pain change | 12 months
  NRS values: with a 0-10 scale, where 0 is no pain and 10 is extreme pain

SECONDARY OUTCOMES:
mood anxiety : zung scale | 12 months
  20-items: score 0 - 44: no anxiety; 45 - 59 moderate anxiety; 60 - 80 severe anxiety

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - AOU Dulbecco Catanzaro, Catanzaro, Italia
  - Luca Gallelli, Catanzaro